CLINICAL TRIAL: NCT00680407
Title: A Multicenter, Randomized, Placebo Controlled Study to Assess the Safety and Efficacy of Orally Administered Silymarin Preparation (Legalon®) for the Treatment of Non-Cirrhotic Patients With Non-Alcoholic Steatohepatitis
Brief Title: Phase II Trial of Silymarin for Non-Cirrhotic Patients With Non-Alcoholic Steatohepatitis
Acronym: SyNCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Madaus Inc (Industry)
Collaborators: University of Pennsylvania (Other); University of North Carolina (Other); Thomas Jefferson University (Other); Beth Israel Deaconess Medical Center (Other); Brooke Army Medical Center (U.S. Federal Agency); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01AT003566-02 (NIH); IND 105,461 (orig. IND 74,887) (Other: FDA Investigational New Drug Application)
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: NASH; non-alcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Lactose; Silymarin; milk-thistle extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- silymarin 420 mg (Experimental): 420 mg Legalon (silymarin) three times daily
  Interventions: Drug: Silymarin 420 mg
- silymarin 700 mg (Experimental): 700 mg of Legalon (silymarin) three times daily
  Interventions: Drug: Silymarin 700 mg
- Placebo (Placebo Comparator): Placebo (lactose pill)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo (5 pills, three times daily) for 48-50 week treatment period
  Other Names: lactose pill
  Arms: Placebo
Drug: Silymarin 700 mg — 700 mg dose (5 pills, three times daily) for 48-50 week treatment period
  Other Names: Legalon; milk thistle
  Arms: silymarin 700 mg
Drug: Silymarin 420 mg — 420 mg dose (5 pills, three times daily) for 48-50 week treatment period
  Other Names: Legalon; milk thistle
  Arms: silymarin 420 mg

SUMMARY:
Silymarin, also known as milk thistle, is an alternative medicine commonly found in health food and vitamin stores. People with liver disease sometimes use silymarin because it is thought to have liver protecting effects; however, this benefit has not been proven. The purpose of this research study is to determine the effectiveness of silymarin and assess the safety of different silymarin doses in patients with varying severity of liver disease compared to a placebo (lactose pill).

Following a screening visit, patients with histologically confirmed NASH will be randomized to either placebo or one of two active treatment groups of silymarin (Legalon®). One active treatment group will receive 420 mg, each dose given three times daily, the other active treatment group will receive 700 mg, each dose given three times daily. Patients will be treated for 48-50 weeks. Participation in this research study requires the patient to travel to the clinic for at least 11 visits so recruitment will be limited to a geographically restricted area around participating clinical centers. Liver biopsy must be performed up to 12 months prior to, and immediately after, the treatment phase.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double masked, placebo controlled Phase II trial to evaluate the safety and explore the efficacy of silymarin (Legalon®) compared with placebo on hepatic histology in patients with NASH (nonalcoholic steatohepatitis) after 48-50 weeks of therapy. This study was originally sponsored through a cooperative agreement (U01) award from the NCCAM and the NIDDK (RFA-AT-05-006: "Phase I/II Trials of Silymarin for Chronic Liver Diseases"), and now will continue with Madaus Inc. (Rottapharm Group) providing financial and regulatory support to the investigators. The broad aim of this study is to evaluate the safety and explore the efficacy of silymarin (Legalon®) in NASH patients and to form the basis for future studies which will establish its efficacy for treating patients with NASH. The specific objectives of this study are to determine the effect of silymarin (Legalon®) on the histologic NASH Activity Score (NAS), the liver enzymes, and HOMAr. The primary endpoint of the study is an improvement in the NAS by at least 2 points. Various secondary endpoints will be assessed, including the change in liver enzymes and HOMAr.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years at screening.
* Informed consent signature.
* AST (aspartate aminotransferase) or ALT (alanine aminotransferase) greater than 40 IU/L within one year of screening and at least once during the screening period.
* The participant must agree to adhere to the alcohol consumption guidelines.
* Have a liver biopsy performed within 12 months of randomization demonstrating features consistent with NASH without cirrhosis; NAS score of at least 4. Historical biopsy must include one Trichrome and one H&E slide, otherwise the biopsy must be redone.
* No change in diabetic medications or insulin sensitizers (if applicable) between biopsy and screening or during the screening period.
* Weight loss/gain of no more than 10% between biopsy and screening, or within 30 days of screening if the biopsy is performed during the screening period.
* Negative urine pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study medication. Females of childbearing potential must be using two reliable forms of effective contraception during the study (while on study drug and during follow-up).

Exclusion Criteria:

* Use of silymarin or other milk thistle preparations for a period of 90 consecutive days or longer between biopsy and initial screening, or within 30 days prior to screening if the biopsy is performed during the screening period.
* Use of other antioxidants such as vitamin E, vitamin C, glutathione, alpha-tocopherol, or non-prescribed complementary alternative medications (including dietary supplements, megadose vitamins, herbal preparations, and special teas) within 30 days prior to screening. A multivitamin at standard doses will be allowed.
* Use of silymarin or other antioxidants or non-prescribed complementary alternative medications (as above) during the screening period or patient unwilling to refrain from taking these medications through completion of the study.
* BMI > 45 kg/m2 between screening and randomization.
* Type 2 diabetes treated with oral agents other than the secretagogues or metformin; these include, thiazolidinediones, alpha-glucosidase inhibitors, exenatide, pramlintide between screening and randomization. Januvia (sitagliptin) is allowed.
* Evidence of poorly-controlled diabetes (defined as HbA1c > 8% in patients with diabetes) between screening and randomization.
* Known allergy/sensitivity to milk thistle or its preparations.
* Use of drugs associated with a clinical or histological picture consistent with fatty liver disease or NASH for more than 12 consecutive weeks in the 1 year prior to screening; these include amiodarone, tamoxifen, methotrexate, glucocorticoids, anabolic steroids, tetracyclines, estrogens at doses greater than those used for hormone replacement, valproate/valproic acid.
* For patients using antihyperlipidemic agents or accepted anti-diabetic agents, any change of agent or dose from screening through randomization.
* Use of warfarin, metronidazole, or acetaminophen (greater than 2 grams per day) from screening through randomization.
* Lactose intolerance defined as patient reported inability to tolerate milk products.
* History of other chronic liver disease, including metabolic diseases, documented by appropriate test(s).
* Previous liver biopsy that demonstrated presence of cirrhosis.
* Radiologic imaging consistent with cirrhosis or portal hypertension.
* Clinical or histological evidence of cirrhosis or, in the opinion of the investigator, the inability to safely obtain a liver biopsy due to technical reasons, such as body habitus.
* Evidence of decompensated liver disease defined as any of the following: serum albumin <3.2 g/dl, total bilirubin > 1.5 mg/dl, or PT/INR (Prothrombin Time/International Normalized Ratio) > 1.3 times normal at screening, or history or presence of ascites or encephalopathy, or bleeding from esophageal varices.
* Platelet count < 130,000/mm3 at screening.
* Serum creatinine of 2.0 mg/dL or greater or CrCl ≤ 60cc/min, or on dialysis, at screening. The creatinine clearance (CrCl) will be calculated according to Cockcroft-Gault.
* Average alcohol consumption of more than one drink or equivalent (>12 grams) per day or more than two (2) drinks on any one day over the 30 days prior to screening. Patients who met either criterion more than 30 days prior to screening must have consumed a monthly average of 12 grams or less per day of alcohol for at least six months prior to screening.
* Evidence of drug abuse in the year prior to screening or prior to randomization.
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, severe psoriasis, rheumatoid arthritis) that could affect the assessment of biomarkers of inflammation.
* History of solid organ or bone marrow transplantation.
* History of thyroid disease poorly controlled on prescribed medications.
* Use of oral steroids for more than 14 days within 30 days of screening or prior to randomization.
* Primary hepatic malignancy.
* Secondary hepatic malignancy (metastatic disease) or extrahepatic malignancy.
* Women with ongoing pregnancy or breast feeding, or contemplating pregnancy.
* History of bariatric surgery, or undergoing evaluation for bariatric surgery.
* Participation in a research drug trial, exclusive of the SyNCH Phase I trial, within 30 days of screening.
* History or other evidence of severe illness or any other conditions that would make the patient, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, coronary artery disease, or active gastrointestinal conditions that might interfere with drug absorption).
* Inability or unwillingness to give informed consent or abide by the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fried, MD, Principal Investigator — University of North Carolina, Chapel Hill; Victor Navarro, MD, Principal Investigator — Thomas Jefferson University; Nezam Afdhal, MD, Principal Investigator — Beth Israel Deaconess Medical Center; K. Rajender Reddy, MD, Principal Investigator — University of Pennsylvania; Steven H. Belle, PhD, Principal Investigator — University of Pittsburgh; Stephen A. Harrison, MD, Principal Investigator — Brooke Army Medical Center
Locations (6):
- United States (6):
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brooke Army Medical Center, San Antonio, Texas

REFERENCES:
- [Derived] Navarro VJ, Belle SH, D'Amato M, Adfhal N, Brunt EM, Fried MW, Reddy KR, Wahed AS, Harrison S; Silymarin in NASH and C Hepatitis (SyNCH) Study Group. Silymarin in non-cirrhotics with non-alcoholic steatohepatitis: A randomized, double-blind, placebo controlled trial. PLoS One. 2019 Sep 19;14(9):e0221683. doi: 10.1371/journal.pone.0221683. eCollection 2019. PMID 31536511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 5 sites; first observation April 30, 2008, last observation Nov 12, 2012.
Period: Overall Study
Arm/Group | Silymarin 420 mg | Silymarin 700 mg | Placebo
Started | 26 | 27 | 25
Completed | 18 | 22 | 22
Not Completed | 8 | 5 | 3
Not completed — Lost to Follow-up | 3 | 3 | 1
Not completed — Withdrawal by Subject | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silymarin 420 mg | Silymarin 700 mg | Placebo | Total
Number analyzed (Participants) | 26 | 27 | 25 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (10.83) | 48.2 (11.43) | 49.51 (10.89) | 48.3 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 11 | 33
  Male | 13 | 18 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - Improvement by at Least 2 Points in Histology (NAS)
Description: Histological Scoring System for Nonalcoholic Fatty Liver Disease ranges from 0-8 with the increase in number representing a worse outcome. Therefore the efficacy improvement was to be at least 2 points in lowering the score.
Time Frame: 48-50 week treatment period
Measure: Number; unit: participants
Arm/Group | Silymarin 420 mg | Silymarin 700 mg | Placebo
Number analyzed (Participants) | 26 | 27 | 25
participants | 5 | 4 | 3

2. Secondary Outcome: Safety - Occurrence of a Dose-limiting Toxicity
Time Frame: 48-50 week treatment period
Measure: Number; unit: participants
Arm/Group | Silymarin 420 mg | Silymarin 700 mg | Placebo
Number analyzed (Participants) | 26 | 27 | 25
participants | 2 | 0 | 0

3. Post Hoc Outcome: Efficacy - Improvement by at Least 2 Points in Histology (NAS) - With NAS Without Cirrhosis
Description: This outcome measure excludes the substantial percentage (62.8%) of patients with baseline biopsies that were deemed ineligible (per inclusion criteria) by the central pathologist due to NAS <4 or absence of NASH (nonalcoholic steatohepatitis) (n=34), NASH with presence of cirrhosis (n=1), or slides unavailable/not evaluable for reading (n=14).
Time Frame: 48-50 week treatment period
Population: Subgroup of ITT (Intent to Treat) Patients with NASH and without cirrhosis population
Measure: Number; unit: participants
Arm/Group | Silymarin 420 mg | Silymarin 700 mg | Placebo
Number analyzed (Participants) | 10 | 9 | 10
participants | 3 | 4 | 1

ADVERSE EVENTS:
Arm/Group | Silymarin 420 mg | Silymarin 700 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/26 | 2/27 | 1/25
Other Adverse Events (participants affected / at risk) | 17/26 | 14/27 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silymarin 420 mg (N=26) | Silymarin 700 mg (N=27) | Placebo (N=25)
ACUTE HEMATOMA POST TREATMENT LIVER BIOPSY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HOSPITALIZED FOR SEVERE HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
LOW PLATELET COUNT (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
BACK SURGERY L5/S1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Silymarin 420 mg (N=26) | Silymarin 700 mg (N=27) | Placebo (N=25)
Gasto-intestinal (Gastrointestinal disorders) | 5 | 4 | 4
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Cardiac (Cardiac disorders) | 3 | 1 | 2
Depression (Nervous system disorders) | 1 | 2 | 1
Dermatologic (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Headache (General disorders) | 2 | 1 | 2
Hyperglycemia (Investigations) | 1 | 2 | 0
Neurological (Psychiatric disorders) | 0 | 1 | 2
Urological (Renal and urinary disorders) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No